CLINICAL TRIAL: NCT01207141
Title: Pharmacodynamics, Pharmacogenomics, and Preliminary Safety and Efficacy of rATG Induction and Tacrolimus Monotherapy in Pediatric Liver Transplantation
Brief Title: rATG Induction and Tacrolimus Monotherapy in Pediatric Liver Transplantation
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rakesh Sindhi, Professor of Surgery, University of Pittsburgh
Other Study IDs: 0608006; 1R01AI073895-01 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Liver Transplantation; Thymoglobulin; Rejection
Keywords: Liver Transplantation; Thymoglobulin; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- rATG induction: Liver transplant recipients who receive induction with rATG prior to transplantation.
- no rATG induction: Liver transplant recipients who do not receive rATG induction therapy prior to transplantation.

SUMMARY:
This open-label clinical trial will evaluate the pharmacodynamics, pharmacogenomics and early efficacy and safety of steroid-free Tacrolimus (TAC) monotherapy and its minimization after induction with rabbit, anti-human thymocyte globulin (rATG, Genzyme, Cambridge, MA) in children and adults with pediatric liver transplantation. Eighty subjects (0-21 years) receiving liver transplantation will be enrolled. Incidence and severity of biopsy-proven acute cellular rejection (ACR) is a primary endpoint as well as time to Tacrolimus whole blood concentrations <8 ng/ml The expected incidence of ACR is 50% and is derived from a non-consecutive subject population (n=40) who received an identical regimen in IND 64555. This incidence is acceptable because the long term sequel of rejection reported with other allografts have not been observed in liver grafts during IND 64555. These risks are further negated by the unique regenerative capacity of the liver allograft. An OBSERVATIONAL arm is being included in this trial. Because the numbers of pediatric liver transplants (LTx) are small in any single center setting, no information is known about relative outcomes on a conventional protocol, in children receiving conventional protocol of steroids+Tacrolimus. The PURPOSE of this additional recruitment is OBSERVATIONAL, only. Therefore, these subjects will NOT be randomized. Rather, by studying all types of patients, the investigators hope to utilize maximally, all available subjects, to understand the relative place of monotherapeutic induction. In turn, this will be the basis for a follow-up comparative, randomized trial.

DETAILED DESCRIPTION:
This open-label clinical trial will evaluate the pharmacodynamics, pharmacogenomics and early efficacy and safety of steroid-free Tacrolimus (TAC) monotherapy and its minimization after induction with rabbit, anti-human thymocyte globulin (rATG, Genzyme, Cambridge, MA) in children and adults with pediatric liver transplantation. Eighty subjects (0-21 years) receiving liver transplantation will be enrolled. Incidence and severity of biopsy-proven acute cellular rejection (ACR) is a primary endpoint as well as time to Tacrolimus whole blood concentrations <8 ng/ml The expected incidence of ACR is 50% and is derived from a non-consecutive subject population (n=40) who received an identical regimen in Investigational New Drug (IND) 64555. This incidence is acceptable because the long term sequel of rejection reported with other allografts have not been observed in liver grafts during IND 64555. These risks are further negated by the unique regenerative capacity of the liver allograft. An OBSERVATIONAL arm is being included in this trial. Because the numbers of pediatric liver transplants (LTx) are small in any single center setting, no information is known about relative outcomes on a conventional protocol, in children receiving conventional protocol of steroids+Tacrolimus. The PURPOSE of this additional recruitment is OBSERVATIONAL, only. Therefore, these subjects will NOT be randomized. Rather, by studying all types of patients, we hope to utilize maximally, all available subjects, to understand the relative place of monotherapeutic induction. In turn, this will be the basis for a follow-up comparative, randomized trial.

The protocol also incorporates a clearly defined schedule to minimize Tacrolimus (TAC) maintenance therapy in each subject, based on presence or absence of early biopsy-proven rejection.

Secondary clinical endpoints are:

3. Time to steroid elimination. 4. Duration of steroid treatment. 5. Steroid-resistant rejection. 6. Cytomegalovirus (CMV) antigenemia (pp5) and CMV disease 7. Epstein-barr virus (EBV) viremia 8. Post-transplant lymphoproliferative disorder (PTLD) 9. Frequency of use of Non-immunosuppressive co-medications - antihypertensives, magnesium and bicarbonate supplements, hypokalemic agents (safety endpoint).

10. Time to first rejection

Secondary pharmacodynamic and pharmacogenomic endpoints are 1. Longitudinal evaluation of peripheral lymphocyte subsets prior to and at 1, 4, and 12 months after liver transplantation. This will establish the pattern of lymphocyte reconstitution after depletion with rATG. 2. Inheritance disequilibrium of 100,000 single nucleotide polymorphisms in the major histocompatibility region. This will entail pre-transplant characterization of these single-nucleotide polymorphisms (SNPs) in all children and their biological parents. Preliminary studies lead us to expect identification of outcome-specific patterns of inheritance of SNPs. Such patterns could be used in future studies to allocate appropriate treatment to children based on predicted risk of rejection. For example, the predicted rejector could receive steroids with rATG+Tacrolimus, while the non-rejector could avoid steroids completely.

Research Design and Methods:

Study type: This is a prospective, open-label, evaluation of steroid-free, induction immunosuppression in children receiving liver transplantation.

Study population: Children 0- 21 years receiving liver transplantation.

Informed consent: This will be obtained by the PI or his physician co-investigators.

Randomization: Not applicable.

Control group: Not applicable

Test group: rATG pretreatment.

1. Premedication with acetaminophen 10 mg/kg orally + diphenhydramine 1 mg/kg intravenously + methylprednisolone 2 mg/kg, intravenously.
2. rATG 5 mg/kg will be initiated prior to liver transplantation, with half the dose infused over at least 4 hours, prior to reperfusion of the liver graft. Total dose to be infused over 24 hours, but no less than 8 hours. If the requisite amount cannot be infused before LTx, it can be continued through the LTx procedure and afterward.

Procedures:

1. Tacrolimus will be initiated at 0.01 mg per kg body weight orally. If biopsy-proven rejection does not occur, Tacrolimus will be titrated to whole blood concentrations:

   Month 1 12-15 ng/ml Months 2-3 8-12 ng/ml Month 4-6 5-8 ng/ml Months 6-12 <5 ng/ml
2. This minimization protocol will be delayed by 3 months if biopsy proven acute cellular rejection occurs. For example, if rejection occurs, Tacrolimus is increased to month 1 levels of 12-15 ng/ml, and steroids added to the regimen. Steroids will be eliminated within 3 months of rejection, and Tacrolimus minimization resumed as described above. These protocols are our standards of care in the event of rejection, whether we use the rATG induction approach with steroid-free Tacrolimus, or Tacrolimus with steroids.
3. Laboratory tests per clinical protocol. The clinical standard of care will be followed in performing post-LTx monitoring labs consisting of complete blood count with differential count, serum sodium, potassium, chloride, bicarbonate, BUN, creatinine and glucose, and liver function tests consisting of Total bilirubin, aspartate alanine transaminase (ALT), aspartate glutamine transaminase (AST), and glutamyl galactosyl transaminase (GGT), and TAC whole blood concentrations. These laboratory tests are performed at least weekly in the first and second months, twice monthly in month 3, and monthly thereafter to the sixth month. The extra 5 ml needed for pharmacodynamic and pharmacogenomic studies is discussed further in items 5 and 6, and in Table 7.
4. Pharmacogenomic studies will consist of characterizing 100,000 SNPs using a SNP array and DNA extracted from 3 ml of whole blood obtained pre-LTx, from each of 80 children.
5. Table 7 (located in . Blood sampling strategy for: pharmacodynamic studies which will measure the lymphocyte subsetsas well as dendritic cells types 1 and 2 are shown in the following table (table 8). Concentration of rATG will also be measured in 0.1 ml human plasma obtained from the same blood sample. Concentration associated with half-maximal depletion of each subset will be determined by pharmacodynamic models based on Hill equations.

   This assay will be carried out in the laboratories of Dr. Rakesh Sindhi at the Rangos Research Center at 530 45th St, Pittsburgh, Pa 15201. Specimens will be stored in the transplant laboratory indefinitely, and will be under the control of the principal investigator, Dr. Rakesh Sindhi. The specimens will be stored to include assigned code numbers and the information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The specimens will be shared with secondary investigators without identifiers.
6. Liver biopsy will be performed per clinical standard of care, to rule out acute cellular rejection. No protocol biopsies will be performed.
7. The treatment of rejection consists of steroids taper per standard of care. This standard includes methylprednisolone, total dose up to 30 mg/kg, or its equivalent. If this occurs, TAC whole blood concentrations will be titrated starting with 12-15 ng/ml during month 1 following the rejection event. Thereafter, the timing of downward titration of TAC concentrations will follow the schema outlined in item 3.
8. Steroid-resistant rejection is defined as biopsy-proven acute cellular rejection not responsive to methylprednisolone or its equivalent.
9. Follow-up for each patient is 12 months.
10. All children will receive standard of care for antiviral and antipneumocystic prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* Age 0-21 years, male and female
* Primary OLTx, Whole/segmental, cadaveric/live, Re-LTx, and LTx in the setting of a previous or simultaneous kidney transplant.
* All children receiving the types of LTx described above, but on conventional immunosuppression, will be enrolled in an observational arm, with the same treatment and monitoring protocols.

Exclusion Criteria:

* Multiorgan transplants (liver-intestine, liver intestine with stomach and other organs)
* Documented non-compliance
* Donor: Age >60, macrovesicular steatosis > 30%, Hepatitis C and B infections defined as anti-HCV antibody positive, and anti-Hepatitis B surface antigen or Hepatitis B core antibody positive, malignancy, cold ischemia time >16 hours
* Children of child-bearing age receive pregnancy testing at the time of transplantation. Pregnancy is a contraindication to liver transplantation and therefore to enrollment in this clinical trial.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 0- 21 years receiving liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2006-08; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of biopsy-proven acute cellular rejection | 90 days

SECONDARY OUTCOMES:
Time to Tacrolimus whole blood concentrations <8 ng/ml | 1 year
Duration of steroid treatment and time to steroid elimination | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sindhi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States